CLINICAL TRIAL: NCT05159635
Title: The Effectiveness of Combining Active Living Programme (ALP) With Home-Use Wearable Technical Aids (WTA) to Promote Community Participation in Young Stroke With Foot Drop Problem- The Pilot Study
Brief Title: Combining Active Living Programme (ALP) With Home-Use Wearable Technical Aids (WTA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kowloon Hospital, Hong Kong (Other)
Collaborators: Kwong Wah Hospital (Other); Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Marko Chan, Senior Occupational Therapist, Kowloon Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KC/KE-17-0187/FR-3
Record Dates: First submitted 2021-08-04; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Stroke; Foot Drop (Acquired)
Keywords: Wearable
MeSH Terms: conditions — Stroke; Peroneal Neuropathies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Living programme and wearable technical aids (Experimental): Active Living programme and wearable technical aids
  Interventions: Device: Active Living programme and wearable technical aids
- Wearable technical aids (Active Comparator): Wearable technical aids
  Interventions: Device: Wearable technical aids

INTERVENTIONS:
Device: Active Living programme and wearable technical aids — attend 6 weeks active living programme and apply wearable technical aids for 8 weeks.
  Arms: Active Living programme and wearable technical aids
Device: Wearable technical aids — apply wearable technical aids for 8 weeks.
  Arms: Wearable technical aids

SUMMARY:
The objective of this study is to evaluate the effectiveness of adopting a home-use Wearable Technical Aids (WTA) with the structured Active Living Program (ALP) to promote community participation in young stroke patients.

DETAILED DESCRIPTION:
Two groups of patients would receive Wearable Technical Aids Training or Wearable Technical Aids Training and structured Active Living Program (ALP) for 8 sessions.

ELIGIBILITY:
Inclusion Criteria:

-diagnosed with foot drop with tibialis anterior muscle strength between 1 to 3- out of 5 in manual muscle testing for more than six months due to cerebrovascular accident (CVA)

Exclusion Criteria:

* pre-existing orthopedic conditions affecting ambulation
* subjects who are incompetent in giving written consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Change score in Stroke Adapted 30 item version of the Sickness Impact Profile (SA-SIP 30) | before intervention, 8 weeks (after intervention )
  The quality of life scale for the people with stroke

SECONDARY OUTCOMES:
Change score in 10 meters walk Test | before intervention,8 weeks (after intervention)
  10 meters walk time

CONTACTS AND LOCATIONS:
Overall Officials: Marko Chan, MSc, Principal Investigator — Community Rehabilitation Service Supoort Centre
Locations (1):
- Community Rehabilitation Service Support Centre, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No